CLINICAL TRIAL: NCT05548634
Title: A 2-Part Open-Label Phase I Study of TAVO412 in Patients with Advanced or Metastatic Solid Tumors Who Progressed on Prior Approved Standard of Care Therapy
Brief Title: A Study of TAVO412 in Patients with Cancer
Acronym: TAVO412
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tavotek Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 59870003
Record Dates: First submitted 2022-09-14; First posted 2022-09-21 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Part 1 Cohort 0 (Other): IV infusion of TAVO412
  Interventions: Drug: TAVO412
- Part 1 Cohort 1 (Other): IV infusion of TAVO412
  Interventions: Drug: TAVO412
- Part 1 Cohort 2 (Other): IV infusion of TAVO412
  Interventions: Drug: TAVO412
- Part 1 Cohort 3 (Other): IV infusion of TAVO412
  Interventions: Drug: TAVO412
- Part 1 Cohort 4 (Other): IV infusion of TAVO412
  Interventions: Drug: TAVO412
- Part 1 Cohort 5 (Other): IV infusion of TAVO412
  Interventions: Drug: TAVO412
- Part 2 Cohorts (Other): IV infusion of TAVO412
  Interventions: Drug: TAVO412

INTERVENTIONS:
Drug: TAVO412 — Biologic

SUMMARY:
TAVO412 Phase 1 is an open-label, non-randomized, 2-part Phase I study to examine the safety, tolerability, pharmacokinetics/pharmacodynamics, and preliminary efficacy of TAVO412. Part 1 will utilize a standard 3 + 3 design to determine the MTD/RP2D of TAVO412 in subjects with advanced or metastatic solid tumors who progressed on prior approved standard of care therapy. Part 2 will further evaluate the safety, tolerability, preliminary efficacy, pharmacokinetics (PK), and pharmacologic activity of TAVO412 in a new set of subjects with advanced or metastatic gastric cancer, non-small cell lung cancer (NSCLC), or subjects of other solid tumor types with best clinical responses (e.g., CR > PR > SD) from Part 1 that progressed on prior approved standard of care therapy.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, Phase I study to determine the safety and tolerability, define the MTD/RP2D, and assess the preliminary efficacy of TAVO412 in subjects with advanced or metastatic solid tumors who progressed on prior approved standard of care therapy. Subjects will receive TAVO412 at the tested dose intravenously on Day 1 and 15 in Cycle 1 and will continue this bi-weekly treatment schedule for all future cycles.

The study will be conducted in 2 parts:

* Part 1 - Dose Escalation will determine the MTD and/or RP2D of TAVO412, which includes defining the optimal dose administration schedule.
* Part 2 - Cohort Expansion will evaluate the recommended dose and administration schedule (MTD/RP2D) determined in Part 1 in a new set of subjects with advanced or metastatic gastric cancer, non-small cell lung cancer (NSCLC), or subjects of other solid tumor types with best clinical responses (e.g., CR > PR > SD) from Part 1 that progressed on prior approved standard of care therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male/Female aged 18 (at the time of screening) or older.
2. Willingness to provide written informed consent for the study.
3. Locally relapsed or refractory disease; locally advanced disease must not be amenable to resection with curative intent.
4. Subjects who have disease progression after treatment with available therapies that are known to confer clinical benefit, or who are intolerant to treatment, or who refuse standard treatment. There is no limit to the number of prior treatment regimens.
5. Presence of measurable disease based on RECIST v1.1. Tumor lesions situated in a previously irradiated area, or in an area subjected to other locoregional therapy, are not considered measurable unless there has been demonstrated progression in the lesion.
6. Part 1: Subjects with advanced or metastatic solid tumors who progressed, or refused, or are considered not eligible, on prior approved standard of care therapy. The following will also apply for Part 2 of the study.

   1. Patients with NSCLC who have sensitizing EGFR mutations must have experienced disease progression on prior EGFR TKIs while those with tumor cMET genomic alterations or over-expression must have received prior anti-PD1 agents and platinum-based chemotherapy either in combination or sequentially.
   2. Patients with gastric cancer or gastroesophageal cancer must have received prior cytotoxic chemotherapy and immune checkpoint inhibitor therapy, and where indicated, also received prior HER2-drected therapy or other FDA-approved targeted therapy.
   3. Patients with colorectal cancer must have received fluoropyrimidine, oxaliplatin, and irinotecan ± VEGF-targeting monoclonal antibodies as prior therapy. Patients with RAS-wild type tumors should have received approved anti-EGFR monoclonal antibody. Patients with MSI-high/dMMR colorectal cancer must have received prior immune checkpoint inhibitor therapy
   4. Patients with TNBC must have experienced disease progression on the following as prior therapies:
   5. Pembrolizumab plus chemotherapy (CPS ≥ 10%)
   6. Sacituzumab
   7. Trastuzumab-deruxtecan (HER2-low)
7. Part 2: A new set of subjects with advanced or metastatic gastric cancer, non-small cell lung cancer (NSCLC), or subjects of other solid tumor types with best clinical responses (e.g., CR > PR > SD) from Part 1 that progressed on prior approved standard of care therapy.

   1. For subjects with Gastric Cancer: histologically confirmed Gastric or Gastro-Esophageal Junction Carcinoma (including adenocarcinoma arising from the lower esophagus). If multiple eligible patients exist, preference will be given to enroll subjects with cMet or EGFR mutations, over-expression, or gene amplification.
   2. For subjects with NSCLC: histologically or cytologically confirmed tumor must be NSCLC with EGFR and/or cMet mutations, over-expression, or gene amplification.
8. Part 2: Willingness to undergo pretreatment and on-treatment tumor biopsies (core or excisional).

   Note: A baseline biopsy obtained for other purposes (i.e., not a protocol-defined procedure) before signing consent may be utilized if the subject has not had any intervening systemic therapy from the time of the biopsy to the start of treatment (i.e., Cycle 1 Day 1), and if a minimum of 20 slides or preferably 1 tissue block can be submitted.

   Note: If a subject is scheduled to have a tumor biopsy for the purposes of this study and it is subsequently determined that tumor tissue cannot safely be obtained, then the subject may still enroll in the study. The subject may be replaced within the cohort.
9. For both Part 1 & Part 2, subjects willing to consent to collection of additional blood or tissue samples for exploratory biomarker or genomic analysis purposes.
10. ECOG performance status 0 or 1.
11. Female subjects of child-bearing potential (defined as women who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy and are not postmenopausal, defined as ≥ 12 months of amenorrhea) must have a negative serum pregnancy test at screening.

    1. All female subjects of child-bearing potential must agree to take appropriate precautions to avoid pregnancy (with at least 99% certainty) from screening through 60 days after the last dose of study drug.
    2. All male subjects must agree to take appropriate precautions to avoid pregnancy with a partner (with at least 99% certainty) from screening through 90 days after the last dose of study drug. Permitted methods that are at least 99% effective in preventing pregnancy (see Appendix A) should be communicated to the subjects and their understanding confirmed.
12. Patients with prior malignancies of the same or different tumor type and patients with concurrent malignancies of the same or different tumor type will be included
13. Patients with mild and moderate hepatic impairment (defined as the equivalent of National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) grade 1 toxicity), as well as those with aspartate transaminase (AST) and alanine transaminase (ALT) elevations defined as grade 3 by the NCI CTCAE (> 5 to 20 x ULN (upper limit of normal)), may be asymptomatic and able to tolerate doses equivalent to patients with normal hepatic function
14. Patients with compromised renal function must meet creatinine clearance ≥ 30 mL/minute (estimated by the Cockcroft-Gault formula, [140 - age] × body weight/plasma creatinine × 72 [× 0.85 if female])
15. Patients with Human Immunodeficiency Virus (HIV)/Hepatitis B (HBV)/Hepatitis C (HBC) will be allowed to enter into the study provided the following criteria are met:

    a) Patients with HIV infection must have CD4+ T-cell (CD4+) counts ≥ 350 cells/µL.
16. The following eligibility criteria are for patients with evidence of chronic HBV infection or patients with history of chronic hepatitis C virus (HCV) or who are virologically suppressed on HCV treatment:

    1. Liver-related laboratory eligibility criteria should be the same as that for the general population.
    2. Exceptions: Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) and bilirubin criteria may be less stringent in patients with cancers such as hepatocellular carcinoma and cholangiocarcinoma in whom hepatic function based on Child-Pugh score should be used.
    3. Patients with chronic HBV infection with active disease who meet the criteria for anti-HBV therapy should be on a suppressive antiviral therapy prior to initiation of cancer therapy.

       Note: Subjects with no prior history of hepatitis B infection who have been vaccinated against hepatitis B and who have a positive antibody against hepatitis B surface antigen test as the only evidence of prior exposure may participate in the study.
    4. Patients on concurrent HCV treatments must have HCV below the limit of quantification.
    5. Patients with untreated HCV may be enrolled if the HCV is stable, the patient is not at risk for hepatic decompensation, and the investigational cancer treatment is not expected to exacerbate the HCV infection.
17. Patients without a history of AIDS-defining opportunistic infections or no opportunistic infection within the past 12 months. With the exception of:

    1. Patients with a history of AIDS-defining cancers (e.g., Kaposi's sarcoma, aggressive B-cell lymphoma, and invasive cervical cancer).
    2. Patients on prophylactic antimicrobials where there may be drug-drug interactions or overlapping toxicities should if appropriate, be changed to an alternative antimicrobial, or if not, be excluded.
18. To ensure that effective antiretroviral therapy is tolerated and that toxicities are not confused with investigational drug toxicities, trial participants should be on established ART for at least four weeks and have an HIV viral load less than 400 copies/mL prior to enrollment. However, exclusion may be based on specific ART drugs with overlapping toxicity.

Exclusion Criteria:

1. Laboratory and medical history parameters not within the protocol-defined range. If the screening laboratory tests below were conducted > 7 days before treatment initiation, they will need to be repeated on Day 1 before initiation of treatment.

   1. Absolute neutrophil count < 1.5 × 109/L.
   2. Platelets < 100 × 109/L.
   3. Hemoglobin < 9 g/dL or < 5.6 mmol/L.
   4. Creatinine clearance < 30 mL/minute (estimated by the Cockcroft-Gault formula, [140 - age] × body weight/plasma creatinine × 72 (× 0.85 if female)
   5. Aspartate aminotransferase, alanine aminotransferase, and alkaline phosphatase ≥ 2.5 × ULN.

      Note: Subjects with 1) bone metastases and 2) no hepatic parenchymal metastases on screening radiographic examinations may enroll if the alkaline phosphatase ≤ 5 × ULN. Subjects with 1) bone metastases and/or 2) hepatic parenchymal metastases on screening radiographic examinations may enroll if the alkaline phosphatase is ≤ 5 × ULN only with medical monitor approval.
   6. Total bilirubin ≥ 1.5 × ULN unless conjugated bilirubin ≤ ULN (note: conjugated bilirubin only needs to be tested if total bilirubin exceeds ULN). If there is no institutional ULN, then direct bilirubin must be < 40% of total bilirubin.
   7. International normalized ratio, prothrombin time, or activated partial thromboplastin time > 1.5 × ULN.
2. Transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including granulocyte colony-stimulating factor, granulocyte macrophage colony- stimulating factor, or recombinant erythropoietin) within 14 days before study Day 1.
3. Receipt of anti-cancer medications or investigational drugs within the following intervals before the first administration of study drug:

   1. ≤ 14 days for chemotherapy, targeted small molecule therapy, or radiation therapy. Subjects must also not require chronic use of corticosteroids and must not have had radiation pneumonitis as a result of treatment. A 1-week washout is permitted for palliative radiation to non-central nervous system (CNS) disease with sponsor approval.

      Note: Bisphosphonates and denosumab are permitted concomitant medications.
   2. ≤ 28 days for prior immunotherapy or persistence of active cellular therapy (i.e., chimeric antigen receptor T-cell therapy; other cellular therapies must be discussed with medical monitor to determine eligibility).
   3. ≤ 28 days for a prior monoclonal antibody used for anticancer therapy with the exception of denosumab.
   4. ≤ 7 days for immune-suppressive-based treatment for any reason. Note: Use of inhaled or topical steroids or corticosteroid use for radiographic procedures is permitted.

      Note: The use of physiologic corticosteroid replacement therapy may be approved after consultation with the medical monitor.
   5. ≤ 28 days or 5 half-lives (whichever is longer) before the first dose for all other investigational agents or devices. For investigational agents with long half-lives (e.g., > 5 days), enrollment before the fifth half-life requires medical monitor approval.
4. Has not recovered to ≤ Grade 1 from toxic effects of prior therapy (including prior immunotherapy) and/or complications from prior surgical intervention before starting therapy.

   Note: Subjects with stable chronic AEs (≤ Grade 2) not expected to resolve (such as neuropathy and alopecia) are exceptions and may enroll with medical monitor approval.

   Note: Subjects with a history of any grade immune-related ocular AEs will be excluded.

   Note: Subjects with a history of a Grade 3 or higher immune-related AE from prior immunotherapies are excluded from the dose escalation portion of the study.
5. Receipt of a live vaccine within 30 days of planned start of study drug. Note: Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox/zoster, yellow fever, rabies, Bacillus Calmette-Guérin, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; COVID booster vaccines are permitted ≥ 4 weeks post; however, intranasal influenza vaccines are live attenuated vaccines and are not allowed.
6. Active autoimmune disease that required systemic treatment in the past (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs).

   Note: Subjects who have not required systemic treatment in the past 2 years should discuss their case with medical monitor to determine eligibility.

   Note: Subjects with hyper/hypothyroidism are eligible to participate. Note: Replacement and symptomatic therapies (e.g., levothyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) are not considered a form of systemic treatment and are allowed.
7. Known active CNS metastases and/or carcinomatous meningitis. Note: Subjects with previously treated brain metastases may participate provided that they are stable (without evidence of progression by imaging for at least 28 days before the first dose of study drug and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases or CNS edema, and have not required steroids for at least 14 days before the first dose of study drug.
8. Evidence of active, noninfectious pneumonitis or history of interstitial lung disease.
9. Active infection requiring systemic therapy, including COVID-19.
10. Known allergy or reaction to any component of study drug or formulation components.
11. Is a female who is pregnant or breast feeding, or expecting to conceive children within the projected duration of the study, starting with the screening visit through 60 days after the last dose of study drug OR;
12. Is a male who is expected to father children within the duration of the study, starting with the screening visit through 90 days after the last dose of study drug.
13. Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the subject; or interfere with interpretation of study.
14. Inability to comprehend or unwillingness to sign the informed consent form (ICF).
15. Subject has a history of class III or IV congestive heart failure or severe nonischemic cardiomyopathy, unstable or poorly controlled angina, myocardial infarction, ventricular arrhythmia, or coronary/peripheral artery bypass graft within the previous 6 months of starting study treatment. Furthermore, subject should have no history of cerebrovascular accident, transient ischemic attack, or symptomatic pulmonary embolism, or uncontrolled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of TAVO412 according to Adverse Events and Number of Participants With Dose Limiting Toxicity (DLT) using National Cancer Institute CTCAE v5.0 | Approximately 12 months
  According to the frequency, duration, and severity of Adverse Events (AEs). The Dose Limiting Toxicity (DLT) is based on drug related adverse events and includes unacceptable hematologic toxicity, non-hematologic toxicity of Grade 3 or higher, or elevations in hepatic enzymes suggestive of drug-induced liver injury.
  The Common Terminology Criteria for Adverse Events (CTCAE) v5.0 has a minimum value of Grade 1, or mild, and a maximum value of Grade 4, Life-threatening; pressor or ventilatory support indicated. All DLTs will be assessed by the investigator using National Cancer Institute CTCAE v5.0.

SECONDARY OUTCOMES:
Maximum Serum Concentration (Cmax) of TAVO412 | Approximately 12 months
  The Cmax is the maximum observed serum concentration of TAVO412.
Time to Reach Maximum Observed Serum Concentration (Tmax) of TAVO412 | Approximately 12 months
  The Tmax is defined as time to reach maximum observed serum concentration of TAVO412.
Minimum Serum Concentration (Cmin) of TAVO412 | Approximately 12 months
  The Cmin is the minimum observed serum concentration of TAVO412.
Area Under the Serum Concentration-Time Curve From 0-1 (AUC[t0-t1]) | Approximately 12 months
  The AUC(t0-t1) is the area under the serum TAVO412 concentration-time curve from time t0 to t1.
Overall Response Rate (ORR) | Approximately 12 months
  ORR is defined as the percentage of subject having complete response (CR) or partial response (PR).
Duration of Response (DOR) | Approximately 12 months
  DOR is defined as the time from earliest date of disease response (CR or PR) until earliest date of disease progression.
Progression-Free Survival (PFS) | Approximately 12 months
  PFS is defined as the time from date of first dose of study drug until the earliest date of disease progression.
Duration of Disease Control (CR, PR, and SD) | Approximately 12 months
  Duration of disease control is defined as the sum of PFS followed by maintenance.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Doroshow, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Tisch Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No